CLINICAL TRIAL: NCT01213121
Title: Exploring Alterations of Central Autonomic Modulation in Patients With Bipolar Depression
Brief Title: Neurophysiologic Changes in Patients With Bipolar Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Seung Chang, Clinical Assistant Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: SNUBH 11-2010-040
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Bipolar Depression
Keywords: bipolar depression; heart rate variability; cardio-respiratory coupling; electroencephalography
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bipolar depression (Experimental): unmedicated patients with bipolar depression receiving quetiapine treatment
  Interventions: Drug: Quetiapine
- Control (No Intervention): healthy controls matched for age, gender, and body mass index

INTERVENTIONS:
Drug: Quetiapine — oral tablet/25-600mg per day/once a day/six weeks
  Other Names: Seroquel
  Arms: bipolar depression

SUMMARY:
* To examine differences in neurophysiologic parameters between unmedicated patients with bipolar depression and healthy controls
* To examine within-subject changes in neurophysiologic parameters in patients with bipolar depression treated with quetiapine

DETAILED DESCRIPTION:
* Alterations of neurophysiologic regulation has been suggested in patients with major depressive disorder or bipolar disorders
* Depressive phase of bipolar disorder shows multi-faceted characteristics different from unipolar depression
* Quetiapine is an atypical antipsychotic licensed for treatment of bipolar depression
* The aim of this study is to investigate the pattern of neurophysiologic dysregulation in bipolar depression and its changes induced by quetiapine treatment

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV bipolar disorder I or II
* Depressive phase
* Drug-naive or drug-free

Exclusion Criteria:

* Serious medical or neurological conditions
* DSM-IV substance-related disorders (within 12 months prior to participation)
* Mentally retarded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | Six weeks
  heart rate variability parameters of time/frequency/complexity domains

SECONDARY OUTCOMES:
Cardio-Respiratory Coupling | Six weeks
  integrative parameters of interaction between neurocardiac dynamics and respiratory rhythm
Electroencephalographic Changes | Six weeks
  Electrical brain activities measured by quantitative electroencephalography
Severity of Mood Symptoms | Six weeks
  * Hamilton Depression Rating Scale
  * Bipolar Depression Rating Scale
  * Young Mania Rating Scale
  * Difficulties in Emotion Regulation Scale
  * Emotion Regulation Questionnaire
Severity of Extrapyramidal Symptom Scale | Six weeks
  Drug-Induced Extrapyramidal Symptom Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jae Seung Chang, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Neuropsychiatry, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Berger S, Boettger MK, Tancer M, Guinjoan SM, Yeragani VK, Bar KJ. Reduced cardio-respiratory coupling indicates suppression of vagal activity in healthy relatives of patients with schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Mar 17;34(2):406-11. doi: 10.1016/j.pnpbp.2010.01.009. Epub 2010 Jan 18. PMID 20083149
- [Background] Bar KJ, Schuhmacher A, Hofels S, Schulz S, Voss A, Yeragani VK, Maier W, Zobel A. Reduced cardio-respiratory coupling after treatment with nortriptyline in contrast to S-citalopram. J Affect Disord. 2010 Dec;127(1-3):266-73. doi: 10.1016/j.jad.2010.05.010. Epub 2010 Jun 9. PMID 20538342
- [Background] Chang JS, Yoo CS, Yi SH, Hong KH, Oh HS, Hwang JY, Kim SG, Ahn YM, Kim YS. Differential pattern of heart rate variability in patients with schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Aug 31;33(6):991-5. doi: 10.1016/j.pnpbp.2009.05.004. Epub 2009 May 7. PMID 19427888
- [Background] Kemp AH, Quintana DS, Gray MA, Felmingham KL, Brown K, Gatt JM. Impact of depression and antidepressant treatment on heart rate variability: a review and meta-analysis. Biol Psychiatry. 2010 Jun 1;67(11):1067-74. doi: 10.1016/j.biopsych.2009.12.012. Epub 2010 Feb 6. PMID 20138254
- [Background] Kemp AH, Gray MA, Silberstein RB, Armstrong SM, Nathan PJ. Augmentation of serotonin enhances pleasant and suppresses unpleasant cortical electrophysiological responses to visual emotional stimuli in humans. Neuroimage. 2004 Jul;22(3):1084-96. doi: 10.1016/j.neuroimage.2004.03.022. PMID 15219580
- See also: Click here for more information about recent updates on bipolar disorder research — http://www.nimh.nih.gov/trials/bipolar-disorder-manic-depressive-illness.shtml